CLINICAL TRIAL: NCT07190677
Title: First-line Therapy With Nivolumab Plus Ipilimumab in Combination With Chemotherapy for Metatastatic Non-small Cell Lung Cancer: an Ambispective, Observational, Italian, Multicenter, Real World Study (NICReWo Trial)
Brief Title: First-line Therapy With Nivolumab Plus Ipilimumab in Combination With Chemotherapy for Metatastatic NSCLC (NICReWo Trial)
Acronym: NICReWo
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Francesco Agustoni, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: NICReWo
Record Dates: First submitted 2025-09-15; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: Nivolumab; Ipilimumab; Real world

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
NICReWo is an Italy-wide, multicenter, observational, ambispective study, designed to collect real-life data during the early post-market authorization approval period of the combination nivolumab plus ipilimumab plus chemotherapy.

Data are retrospectively collected starting from January 2022 and will be prospectively collected until 31 December 2025, co-primary endpoints are to evaluate progression-free survival (PFS) and overall survival (OS) in a real world patient population. Secondary endpoints are overall response rate (ORR), duration of treatment and incidence of treatment-related adverse events (AEs). All data obtained for this study are recorded with an Electronic Data Capture (EDC) system using eCRFs (RedCap platform).

DETAILED DESCRIPTION:
The major parameters collected are: patient characteristics (age, sex, ECOG, performance status, smoking status, comorbidities), disease characteristics (NSCLC histology, metastatic sites, molecular profile), treatment timeline (date of starting therapy, number of administered cycles, date and reason of end of therapy, best response, subsequent therapies after disease progression), survival outcomes [PFS (defined as the time from the starting therapy to disease progression or death from any cause) and OS (defined as the time from the starting therapy to death from any cause)]. Data about adverse drug reactions are collected according to the Common Terminology Criteria Adverse Events v5.0. Data collection includes patients treated starting from January 2022 until December, 31 2025, with a 2-years period of follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV or recurrent NSCLC (histologically or cytologically confirmed stage);
* Decision to initiate a first-line treatment with nivolumab plus ipilimumab in combination with 2 cycles of platinum-based chemotherapy for the treatment of NSCLC according to the Italian label, independently of the study, in patients whose tumors have no sensitising EGFR mutation or ALK translocation;
* Patient is at least 18 years of age at time of treatment decision;
* Patient provided written informed consent to participate in the study.

Exclusion Criteria:

* Current primary diagnosis of a cancer other than NSCLC that requires systemic or other treatment;
* Previous treatment with nivolumab and/or ipilimumab;
* Patient already included in an interventional clinical trial for their advanced or recurrent NSCLC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage IV or recurrent NSCLC treated with nivolumab plus ipilimumab in combination with 2 cycles of platinum-based chemotherapy, according to local clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
to estimate OS and PFS | January 2022 - December 2025
  to estimate the overall OS and the PFS after 24 months from start of therapy among patients with stage IV or recurrent NSCLC treated with nivolumab plus ipilimumab in combination with 2 cycles of platinum-based chemotherapy

SECONDARY OUTCOMES:
to estimate OS and PFS under real-life conditions in Italy considering subgroups | January 2022 - December 2025
  To estimate OS and PFS according to subgroups of interest: - ECOG Performance Status (PS): ECOG PS 0-1 and 2; - Presence of brain metastases; - Mediastinal lymph nodes staging: N0, N1, N2, N3; - Presence of extra-thoracic lymph node metastases; - Age >75 years; - Pre-existing autoimmune disorders; - Development of immune-related adverse events (AEs); - PD-L1 negative status; - Genetic mutations and co-mutations (KRAS, MET, BRAF or ROS1 genes or with resistance-conferring mutations in the STK11, KEAP1 and TP53 genes)
to evaluate overall response rates by histology type, other subgroups of interest and treatment characteristics | January 2022 - December 2025
  To estimate the intermediate endpoints of response rates overall and according to histology types, other subgroups of interest and treatment characteristics with 24 months from start of therapy: - Overall response rate [ORR = Complete Response + Partial Response]; - Best overall response rate [BORR]
to assess the overall duration of treatment and subdivide it according to histology types and other subgroups of interest | January 2022 - December 2025
  To estimate duration of treatment overall and according to histology types and other subgroups of interest
to understand the safety of treatment by examining the frequency and severity of adverse events and identifying toxicity | January 2022 - December 2025
  To describe the frequency, severity, and management of following types of adverse events (AEs) to estimate toxicity up to 24 months from start of therapy:
  * Selected immune-related AEs (immune-related pneumonitis, colitis, hepatitis, nephritis/renal dysfunction, endocrinopathies, and rash);
  * Other immune-related AEs (severe infusion reactions, uveitis, pancreatitis, demyelination, Guillain-Barre Syndrome, myasthenic syndrome, encephalitis, toxic epidermal necrolysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy